CLINICAL TRIAL: NCT02974868
Title: A PHASE 2A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTICENTER STUDY TO EVALUATE THE EFFICACY AND SAFETY PROFILE OF PF-06651600 AND PF-06700841 IN SUBJECTS WITH MODERATE TO SEVERE ALOPECIA AREATA WITH A SINGLE-BLIND EXTENSION PERIOD AND A CROSS-OVER OPEN LABEL EXTENSION PERIOD
Brief Title: Study To Evaluate The Efficacy And Safety Profile Of PF-06651600 And PF-06700841 In Subjects With Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Triple | Purpose: Treatment
Other Study IDs: B7931005; 2016-004048-13 (EudraCT Number); ALLEGRO (Other: Alias Study Number)
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Alopecia Areata
Keywords: Phase 2; randomized; double-blind; placebo; alopecia areata; safety; efficacy; JAK; janus kinase; moderate; severe
MeSH Terms: conditions — Alopecia Areata; Lymphoma, Follicular | interventions — PF-06651600; PF-06700841

STUDY DESIGN:
Intervention Model Description: The first 24 weeks are parallel. The single-blind extension period will have a segment for non-responder and a withdrawal/retreatment segment for responder. The cross-over extension period is parallel for non-responders.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): PF-06651600
  Interventions: Drug: PF-06651600
- Cohort 2 (Experimental): PF-06700841
  Interventions: Drug: PF-06700841
- Cohort placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06651600 — 200 mg QD during induction and 50 mg QD during Maintenance
  Arms: Cohort 1
Drug: PF-06700841 — 60 mg QD during induction and 30 mg QD during maintenance
  Arms: Cohort 2
Drug: Placebo — Placebo
  Arms: Cohort placebo

SUMMARY:
This is a Phase 2a, randomized, double blind, parallel group, multicenter study with an extension period. The study will have a maximum duration of approximately 113 weeks. This includes an up to 5 weeks Screening Period, a 24 week Treatment Period, a 4 week Drug Holiday (#1), an up to 12 month Single Blind (investigator open, sponsor open and subject blind) Extension Period, a 4 week drug holiday (#2), a 6 month Cross Over Open Label Extension Period and a 4 week Follow up Period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 75 years of age, inclusive, at time of informed consent.
* Must have moderate to severe alopecia areata:

Exclusion Criteria:

* History of human immunodeficiency virus (HIV) or positive HIV serology at screening,
* Infected with hepatitis B or hepatitis C viruses.
* Have evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB)
* Have received any of the following treatment regiments specified in the timeframes outlined below:

Within 6 months of first dose of study drug: Any cell depleting agents Within 12 weeks of first dose of study drug: Any studies with JAK inhibitors; Other biologics Within 8 weeks of first dose of study drug: Participation in other studies involving investigational drug(s) Within 6 weeks of first dose of study drug: Have been vaccinated with live or attenuated live vaccine.

Within 4 weeks of first dose of study drug: Use of oral immune suppressants; Phototherapy (NB UVB) or broad band phototherapy; Regular use (more than 2 visits per week) of a tanning booth/parlor.

Within 2 week of first dose of study drug: Topical treatments that could affect AA; Herbal medications with unknown properties or known beneficial effects for AA.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (55):
- United States (39):
  - University of Alabama at Birmingham, Dermatology at the Whitaker Clinic, Birmingham, Alabama
  - University of Alabama at Birmingham, The Kirklin Clinic, Birmingham, Alabama
  - Southern California Dermatology, Inc., Santa Ana, California
  - Clinical Science Institute, Santa Monica, California
  - Office of F. Monte Purcelli, Santa Monica, California
  - Tower Saint John's Imaging, Santa Monica, California
  - University of Colorado Hospital Clinical and Translational Research Center, Inpatient Unit, Aurora, Colorado
  - University of Colorado Hospital Clinical and Translational Research Center, Outpatient Clinic, Aurora, Colorado
  - University of Colorado Hospital, Anschutz Cancer Pavilion, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Investigational Drug Services, New Haven, Connecticut
  - Church Street Research Unit, New Haven, Connecticut
  - Yale Hearing and Balance Center, New Haven, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Park Avenue Dermatology Administrative Annex, Orange Park, Florida
  - Park Avenue Dermatology, Orange Park, Florida
  - Edward B. Kampsen, MD, Tampa, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Rose Radiology, Tampa, Florida
  - Forward Clinical Trials, Inc, Tampa, Florida
  - MedaPhase Inc., Newnan, Georgia
  - NorthShore University HealthSystem Dermatology Clinical Trials Unit, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Dawes Fretzin Dermatology Group, LLC, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Clinical Unit for Research Trials in Skin (CURTIS), Boston, Massachusetts
  - Weill Cornell Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Mount Sinai Department of Otolaryngology, New York, New York
  - Rockefeller University Hospital, New York, New York
  - Investigational Drug Service, Rochester, New York
  - University of Rochester Audiology, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of Rochester Radiology, Rochester, New York
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Health Concepts, Rapid City, South Dakota
  - University of Utah MidValley Dermatology, Murray, Utah
  - University of Utah Medical Center, Salt Lake City, Utah
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Australia (10):
  - Hearing Life, Hurstville, New South Wales
  - Dr. Glen and Partners Medical Imaging, Kogarah, New South Wales
  - St George Dermatology and Skin Cancer Centre, Kogarah, New South Wales
  - St. George Hearing and Balance Clinic, Kogarah, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Skin & Cancer Foundation Inc., Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - Bridge Road Imag ing, Richmond, Victoria
  - Richmond Audiology, Richmond, Victoria
- Canada (6):
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Lynderm Research Inc., Markham, Ontario
  - Research by ICLS, Oakville, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - York Dermatology Center, Richmond Hill, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Xi L, Peeva E, Yamaguchi Y, Ye Z, Lejeune A, Hyde C, Guttman-Yassky E. Multiomics Analysis of the Response to Ritlecitinib in Alopecia Areata Subtypes and Correlation With Efficacy. Allergy. 2025 Aug;80(8):2348-2360. doi: 10.1111/all.16659. Epub 2025 Jul 14. PMID 40654284
- [Derived] King B, Soung J, Tziotzios C, Rudnicka L, Joly P, Gooderham M, Sinclair R, Mesinkovska NA, Paul C, Gong Y, Anway SD, Tran H, Wolk R, Zwillich SH, Lejeune A. Integrated Safety Analysis of Ritlecitinib, an Oral JAK3/TEC Family Kinase Inhibitor, for the Treatment of Alopecia Areata from the ALLEGRO Clinical Trial Program. Am J Clin Dermatol. 2024 Mar;25(2):299-314. doi: 10.1007/s40257-024-00846-3. Epub 2024 Jan 23. PMID 38263353
- [Derived] Wojciechowski J, S Purohit V, Huh Y, Banfield C, Nicholas T. Evolution of Ritlecitinib Population Pharmacokinetic Models During Clinical Drug Development. Clin Pharmacokinet. 2023 Dec;62(12):1765-1779. doi: 10.1007/s40262-023-01318-3. Epub 2023 Nov 2. PMID 37917289
- [Derived] Hughes JH, Qiu R, Banfield C, Dowty ME, Nicholas T. Population Pharmacokinetics of Oral Brepocitinib in Healthy Volunteers and Patients. Clin Pharmacol Drug Dev. 2022 Dec;11(12):1447-1456. doi: 10.1002/cpdd.1163. Epub 2022 Aug 31. PMID 36045513
- [Derived] Peeva E, Guttman-Yassky E, Banerjee A, Sinclair R, Cox LA, Zhu L, Zhu H, Vincent M, King B. Maintenance, withdrawal, and re-treatment with ritlecitinib and brepocitinib in patients with alopecia areata in a single-blind extension of a phase 2a randomized clinical trial. J Am Acad Dermatol. 2022 Aug;87(2):390-393. doi: 10.1016/j.jaad.2021.12.008. Epub 2021 Dec 13. No abstract available. PMID 34915057
- [Derived] Guttman-Yassky E, Pavel AB, Diaz A, Zhang N, Del Duca E, Estrada Y, King B, Banerjee A, Banfield C, Cox LA, Dowty ME, Page K, Vincent MS, Zhang W, Zhu L, Peeva E. Ritlecitinib and brepocitinib demonstrate significant improvement in scalp alopecia areata biomarkers. J Allergy Clin Immunol. 2022 Apr;149(4):1318-1328. doi: 10.1016/j.jaci.2021.10.036. Epub 2021 Dec 1. PMID 34863853
- [Derived] Fensome A, Ambler CM, Arnold E, Banker ME, Brown MF, Chrencik J, Clark JD, Dowty ME, Efremov IV, Flick A, Gerstenberger BS, Gopalsamy A, Hayward MM, Hegen M, Hollingshead BD, Jussif J, Knafels JD, Limburg DC, Lin D, Lin TH, Pierce BS, Saiah E, Sharma R, Symanowicz PT, Telliez JB, Trujillo JI, Vajdos FF, Vincent F, Wan ZK, Xing L, Yang X, Yang X, Zhang L. Dual Inhibition of TYK2 and JAK1 for the Treatment of Autoimmune Diseases: Discovery of (( S)-2,2-Difluorocyclopropyl)((1 R,5 S)-3-(2-((1-methyl-1 H-pyrazol-4-yl)amino)pyrimidin-4-yl)-3,8-diazabicyclo[3.2.1]octan-8-yl)methanone (PF-06700841). J Med Chem. 2018 Oct 11;61(19):8597-8612. doi: 10.1021/acs.jmedchem.8b00917. Epub 2018 Aug 16. PMID 30113844
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7931005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study had a 24 week Treatment Period, a 4 week Drug Holiday, an up to 48 weeks(24 weeks + additional 24 Weeks for those received active retreatment) Single Blind Extension Period, a 4 week Drug Holiday, a 24 weeks Cross Over Open Label Extension Period.
Pre-assignment Details: Criteria for entering SBE: complete the former period without showing Key Exclusion defined in CSR Section 9.3.2.
  Criteria for entering COE: non-responders (SALT change from baseline <30%) at Week 24 and continued to be non-responders at Week 52 in SBE period without showing Key Exclusion defined in CSR Section 9.3.2.
Groups:
- Placebo for PF-06651600: Participants received placebo tablets QD matching for PF-06651600.
- Placebo for PF-06700841: Participants received placebo tablets QD matching for PF-06700841.
- PF-06651600: Participants received PF-06651600 200 mg QD for 4 weeks induction period followed by PF-06651600 50 mg QD for a 20 weeks maintenance period.
- PF-06700841: Participants received PF-06700841 60 mg tablets QD for a 4-week induction period followed by PF-06700841 30 mg tablets QD for a 20-week maintenance period.
Period: Initial 24-Week Treatment Period (TP)
Arm/Group | Placebo for PF-06651600 | Placebo for PF-06700841 | PF-06651600 | PF-06700841
Started | 24 | 23 | 48 | 47
Completed | 20 | 14 | 45 | 35
Not Completed | 4 | 9 | 3 | 12
Not completed — Adverse Event | 1 | 1 | 2 | 4
Not completed — others | 3 | 8 | 1 | 8
Period: Single-Blind Extension (SBE) Period
Arm/Group | Placebo for PF-06651600 | Placebo for PF-06700841 | PF-06651600 | PF-06700841
Started (Among 114 participants completed initial treatment period, 96 participants entered SBE period) | 17 | 12 | 38 | 29
Completed (Week 28-52 and additional 24 weeks(AT Day 1 -AT Week 24) for those retreated with active treatment) | 15 | 11 | 27 | 23
Not Completed | 2 | 1 | 11 | 6
Not completed — AE & Withdraw by participants | 2 | 1 | 11 | 6
Period: Cross-Over Extension (COE) Period
Arm/Group | Placebo for PF-06651600 | Placebo for PF-06700841 | PF-06651600 | PF-06700841
Started (Among 76 participants completed SBE period, 23 participants entered COE period.) | 7 | 2 | 11 | 3
Completed (Participants who were PF-06651600 non-responders at Week 52 received PF-06700841, vice versa.) | 5 | 1 | 8 | 3
Not Completed | 2 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: All participants received at least 1 dose of PF-06651600,PF-06700841 or matching placebo.
Groups:
- TP:Placebo: Participants received placebo tablets QD both matching for PF-06651600 and PF-06700841.
- TP:PF-06651600: Participants received PF-06651600 200 mg tablets QD for a 4-week induction period followed by PF-06651600 50 mg tablets QD for a 20-week maintenance period.
- TP:PF-06700841: Participants received PF-06700841 60 mg tablets QD for a 4-week induction period followed by PF-06700841 30 mg tablets QD for a 20-week maintenance period.
- Total: Total of all reporting groups
Arm/Group | TP:Placebo | TP:PF-06651600 | TP:PF-06700841 | Total
Number analyzed (Participants) | 47 | 48 | 47 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.17 (14.22) | 36.88 (12.62) | 33.94 (11.43) | 36.33 (12.84)
Age, Customized [Count of Participants; unit: Participants]
  18-44 Years | 31 | 33 | 40 | 104
  45-64 Years | 15 | 14 | 6 | 35
  >=65 Years | 1 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 37 | 32 | 98
  Male | 18 | 11 | 15 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5 | 10
  Not Hispanic or Latino | 45 | 45 | 42 | 132
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 45 | 38 | 36 | 119
  Black or African American | 0 | 4 | 3 | 7
  Asian | 2 | 3 | 3 | 8
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  other | 0 | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Severity of Alopecia Tool (SALT) Score at Week 24
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. Score range: 0-100%. Higher score indicates more severe disease. Change from baseline is defined as the baseline value minus the value at a specific visit. Positive change from baseline signifies an improvement. Baseline is defined as the last measurement prior to first dosing (Day 1).
Time Frame: Baseline, Week24
Population: Number of Participants Analyzed: All randomized participants assigned to the study treatment. Number Analyzed: Number of Participants with observed data at Week 24
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Groups:
- Placebo: Participants received placebo tablets QD both matching for PF-06651600 and PF-06700841
Arm/Group | PF-06651600 | PF-06700841 | Placebo
Number analyzed (Participants) | 48 | 47 | 47
units on a scale | 32.54 [25.35 to 39.74] | 50.59 [43.15 to 58.02] | 1.41 [-6.03 to 8.85]
Statistical Analysis 1: Comparison: PF-06651600 vs Placebo; Test type: Superiority; p < .0001, Mixed Model Repeated Measure (MMRM) — Hochberg P-value (one-sided); MMRM contains fixed factors of treatment, week, baseline, treatment by week and treatment by baseline interaction and a random effect for subject; Mean of Difference from Placebo = 31.14, 95% CI 2-sided [18.78 to 43.50], Standard Error of Mean 6.25
Statistical Analysis 2: Comparison: PF-06700841 vs Placebo; Test type: Superiority; p < .0001, Mixed Model Repeated Measure (MMRM) — Hochberg P-value (one-sided); [statistical method as in outcome 1, analysis 1]; Mean of Difference from Placebo = 49.18, 95% CI 2-sided [36.62 to 61.74], Standard Error of Mean 6.35

2. Secondary Outcome: Change From Baseline in Severity of Alopecia Tool (SALT) Score at Week 24 -AT/AU Participants
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. The SALT score can vary from 0 to 100%, with higher scores representing increasing severity of disease. Change from baseline is defined as the baseline value minus the value at a specific visit. Positive change from baseline implies an improvement. Alopecia totalis (AT): derived as SALT score = 100% at baseline only. Alopecia universalis (AU): derived as SALT score = 100% and both eyelash and eyebrow assessments were "none" at baseline.
Time Frame: Baseline, Week 24
Population: Number of Participants Analyzed: AT/AU participants in the Full analysis set (FAS) was used. FAS consisted of all randomized participants, assigned to the randomized treatment regardless of what treatment, if any, was received. Number Analyzed: Number of participants with observed data at Week 24.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Groups:
- PF-06651600-AT/AU: AT/AU Participants received PF-06651600 200 mg once daily (QD) for 4 weeks induction period followed by PF-06651600 50 mg QD for a 20 weeks maintenance period.
- PF-06700841-AT/AU: AT/AU Participants received PF-06700841 60 mg tablets QD for a 4-week induction period followed by PF-06700841 30 mg tablets QD for a 20-week maintenance period.
- Placebo-AT/AU: AT/AU Participants received placebo tablets QD both matching for PF-06651600 and PF-06700841.
Arm/Group | PF-06651600-AT/AU | PF-06700841-AT/AU | Placebo-AT/AU
Number analyzed (Participants) | 20 | 22 | 20
units on a scale | 27.59 [15.24 to 39.94] | 48.42 [36.38 to 60.47] | 1.81 [-11.00 to 14.63]
Statistical Analysis 1: Comparison: PF-06651600-AT/AU vs Placebo-AT/AU; Test type: Other; p = 0.0094, Mixed Model Repeated Measure (MMRM); [statistical method as in outcome 1, analysis 1]; Mean of Difference from Placebo = 25.78, 90% CI 2-sided [7.98 to 43.58], Standard Error of Mean 10.64
Statistical Analysis 2: Comparison: PF-06700841-AT/AU vs Placebo-AT/AU; Test type: Other; p < .0001, Mixed Model Repeated Measure; [statistical method as in outcome 1, analysis 1]; Mean of Difference from Placebo = 46.61, 90% CI 2-sided [29.02 to 64.20], Standard Error of Mean 10.51

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (All-causality and Treatment-related) - Single-Blind Extension (SBE) Period
Description: An AE (non-serious and serious) was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Any such events with initial onset or increasing in severity after the first dose of study treatment were counted as treatment-emergent Adverse Event (TEAE). Treatment-related TEAE were determined by investigators. Arms end with "withdrawal Segment" and "retreatment segment" described the same population while in different treatment segment .The reason why count on PF-06700841 differ by 1 participant is that 1 responder directly entered the retreatment segment and skipped the withdrawal segment.
Time Frame: Week 28 up to Week 52
Population: The safety analysis set (SAS) was used , which was defined as all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Active Non-responders on PF-06651600: Participants initially treated with PF-06651600 in the Initial 24-Week Treatment Period and not responsive at Week 24 (ie, not achieving ≥30% improvement from baseline in SALT [SALT 30]) who were continually assigned to PF-06651600 in the Non-Responder Segment of the SBE Period
- Placebo Non-responders on PF-06651600: Participants initially treated with placebo in the Initial 24-Week Treatment Period (1 participant receiving placebo in the Initial 24-Week Treatment Period was responsive at Week 24 but did not enter the SBE Period) who were assigned to PF-06651600 in the Non-Responder Segment of the SBE Period
- Active Non-responders on PF-06700841: Participants initially treated with PF-06700841 in the Initial 24-Week Treatment Period and not responsive at Week 24 (ie, not achieving SALT 30) who were continually assigned to PF-06700841 in the Non-Responder Segment of the SBE Period
- Placebo Non-responders on PF-06700841: Participants initially treated with placebo in the Initial 24-Week Treatment Period who were assigned to PF-06700841 in the Non-Responder Segment of the SBE Period
- Non-Retreated PF-06651600 Responders in the Withdrawal Segment: Participants initially treated with PF-06651600 in the Initial 24-Week Treatment Period and responsive at Week 24 (ie, achieving SALT 30) who were assigned to placebo (withdrawal) without entering the Retreatment Segment of the SBE Period
- Retreated PF-06651600 Responders in the Withdrawal Segment: Participants initially treated with PF-06651600 in the Initial 24-Week Treatment Period and responsive at Week 24 (ie, achieving SALT 30) who were assigned to placebo (withdrawal), and then entered the Retreatment Segment of the SBE Period to receive PF-06651600. This arm stands for retreated responders with TEAE within withdrawal Segment
- Non-Retreated PF-06700841 Responders in the Withdrawal Segment: Participants initially treated with PF-06700841 in the Initial 24-Week Treatment Period and responsive at Week 24 (ie, achieving SALT 30) who were assigned to placebo (withdrawal) without entering the Retreatment Segment of the SBE Period
- Retreated PF-06700841 Responders in the Withdrawal Segment: Participants initially treated with PF-06700841 in the Initial 24-Week Treatment Period and responsive at Week 24 (ie, achieving SALT 30) who were assigned to placebo (withdrawal), and then entered the Retreatment Segment of the SBE Period to receive PF-06700841. This arm stands for retreated responders with TEAE within withdrawal Segment
- Retreated PF-06651600 Responders in the Retreatment Segment: Participants initially treated with PF-06651600 in the Initial 24-Week Treatment Period and responsive at Week 24 (ie, achieving SALT 30) who were assigned to placebo (withdrawal), and then entered the Retreatment Segment of the SBE Period to receive PF-06651600
- Retreated Responders on PF-06700841 in the Retreatment Segment: Participants initially treated with PF-06700841 in the Initial 24-Week Treatment Period and responsive at Week 24 (ie, achieving SALT 30) who were assigned to placebo (withdrawal), and then entered the Retreatment Segment of the SBE Period to receive PF-06700841
Arm/Group | Active Non-responders on PF-06651600 | Placebo Non-responders on PF-06651600 | Active Non-responders on PF-06700841 | Placebo Non-responders on PF-06700841 | Non-Retreated PF-06651600 Responders in the Withdrawal Segment | Retreated PF-06651600 Responders in the Withdrawal Segment | Non-Retreated PF-06700841 Responders in the Withdrawal Segment | Retreated PF-06700841 Responders in the Withdrawal Segment | Retreated PF-06651600 Responders in the Retreatment Segment | Retreated Responders on PF-06700841 in the Retreatment Segment
Number analyzed (Participants) | 16 | 17 | 5 | 12 | 8 | 14 | 9 | 14 | 14 | 15
Participants
  TEAE (All Causalities) | 8 | 12 | 4 | 10 | 4 | 3 | 6 | 9 | 11 | 9
  TEAE (Treatment Related) | 5 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 2

4. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (All-causality and Treatment-related) - Cross-Over Extension (COE) Period
Description: An AE (non-serious and serious) was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Any such events with initial onset or increasing in severity after the first dose of study treatment were counted as treatment-emergent Adverse Event (TEAE). Treatment-related TEAE were determined by investigators.
Time Frame: COE day 1 up to end of study
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- COE-PF-06651600: Participants not responsive to placebo or PF-06700841 at Week 24 in the Initial 24-Week Treatment Period and not responsive to PF-06700841 at Week 52 (ie, not achieving SALT 30) in the SBE Period who were assigned to PF-06651600 in the COE Period
- COE-PF-06700841: Participants not responsive to placebo or PF-06651600 at Week 24 in the Initial 24-Week Treatment Period and not responsive to PF-06651600 at Week 52 (ie, not achieving SALT 30; except 1 PF-06651600 responder) in the SBE Period who were assigned to PF-06700841 in the COE Period
Arm/Group | COE-PF-06651600 | COE-PF-06700841
Number analyzed (Participants) | 5 | 18
Participants
  TEAE (All Causalities) | 4 | 9
  TEAE (Treatment Related) | 2 | 3

5. Primary Outcome: Number of Participants With Laboratory Abnormalities During SBE Period
Description: Following laboratory parameters were assessed against pre-defined abnormality criteria: hematology(Hemoglobin, Hematocrit, RBC count, Reticulocyte count, Platelet count, WBC count with differential, Total neutrophils, Eosinophils, Monocytes, Basophils, Lymphocytes); serum chemistry (BUN and Creatinine, Cystatin C, Creatine Phosphokinase, Glucose , Na+, K+, Cl ,Ca++, Total CO2, AST, ALT, Total Indirect & Direct Bilirubin, Alkaline phosphatase, Uric acid, Albumin,Total protein, Fasting lipid Profile Panel; urinalysis(pH, Glucose, Protein, Nitrites, Leukocyte esterase, Microscopy culture);Other(HIV, HBsAg, HBcAb, HepB reflex (HbsAB), if applicable, HCVAb, Serum pregnancy test, Urine pregnancy test, FSH, QFT G or other IGRA, or PPD, EBV, CMV, HSV1, HSV2, VZV, Skin swab for herpetiform rash, Skin swab for potential drug related rash).Retest/discontinuation criteria are defined in Protocol Appendix 6.1 and 6.2 respectively.
Time Frame: Week 28 up to Week 52 for non-responders and responders in the withdrawal segment, AT day 1 up to AT Week 24 for retreatment segment (AT=active treatment)
Population: The safety analysis set (SAS) was used. Arms end with "withdrawal Segment" and "retreatment segment" described the same population while in different treatment segment .The reason why count on PF-06700841 differ by 1 participant is that 1 responder skipped the withdrawal segment and entered the retreatment segment.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Non-responders on PF-06651600 | Placebo Non-responders on PF-06651600 | Active Non-responders on PF-06700841 | Placebo Non-responders on PF-06700841 | Non-Retreated PF-06651600 Responders in the Withdrawal Segment | Retreated PF-06651600 Responders in the Withdrawal Segment | Non-Retreated PF-06700841 Responders in the Withdrawal Segment | Retreated PF-06700841 Responders in the Withdrawal Segment | Retreated PF-06651600 Responders in the Retreatment Segment | Retreated Responders on PF-06700841 in the Retreatment Segment
Number analyzed (Participants) | 16 | 17 | 5 | 12 | 8 | 14 | 9 | 14 | 14 | 15
Participants
  With abnormalities without regard to baseline | 13 | 11 | 4 | 11 | 6 | 9 | 7 | 10 | 11 | 14
  Meeting Retest Criteria | 3 | 5 | 2 | 7 | 2 | 0 | 3 | 2 | 4 | 4
  Meeting Discontinuation Criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

6. Primary Outcome: Numbers of Participants With Specific Clinical Laboratory Abnormalities During COE Period
Description: as for outcome 5
Time Frame: COE day 1 up to end of study
Population: All participants in safety analysis set (SAS) who received at least 1 dose of investigational product (PF-06651600, PF-06700841 or placebo) and had abnormal laboratory data in COE period.
Measure: Count of Participants; unit: Participants
Arm/Group | COE-PF-06651600 | COE-PF-06700841
Number analyzed (Participants) | 5 | 18
Participants
  With abnormalities without regard to baseline | 5 | 11
  Meeting Retest Criteria | 1 | 6
  Meeting Discontinuation Criteria | 0 | 0

7. Secondary Outcome: Percentage of Participants Achieving SALT 30 at Week 24
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. A SALT 30 response is a 30% or greater reduction from baseline in SALT score. The SALT score can vary from 0 to 100%, with higher scores representing increasing severity of disease. The analysis was done using FAS (full analysis set) based on Non-responder imputation (ie. set missing values to be non-responsive) data. The 90% CI was calculated using Chan and Zhang method.
Time Frame: Baseline, Week 24
Population: All participants in the Full analysis set (FAS) was used and have observed data at Week 24. FAS consisted of all randomized participants, assigned to the randomized treatment regardless of what treatment, if any, was received.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06651600 | PF-06700841 | Placebo
Number analyzed (Participants) | 48 | 47 | 47
percentage of participants | 50.0 [37.6 to 62.4] | 63.8 [51.3 to 74.9] | 2.1 [0.2 to 8.8]
Statistical Analysis 1: Comparison: PF-06651600 vs Placebo; Test type: Other; p < .0001, Chan and Zhang method; Difference in Percentage from Placebo = 47.9, 90% CI 2-sided [34.2 to 60.7]
Statistical Analysis 2: Comparison: PF-06700841 vs Placebo; Test type: Other; p < .0001, Chan and Zhang method; Difference in Percentage from Placebo = 61.7, 90% CI 2-sided [48.2 to 73.6]

8. Secondary Outcome: Change From Baseline in Severity of Alopecia Tool (SALT) Across Time (Treatment Period)
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. The SALT score can vary from 0 to 100% with higher score indicates more severe disease. Baseline is defined as the last measurement prior to first dosing (Day 1). Change from baseline is defined as the baseline value minus the value at a specific visit. Positive change from baseline implies an improvement. Least Square Mean and 90% Confidence Interval of Arms (PF-06651600 and PF-06700841) are the Least Square Mean and 90% Confidence Interval for difference from placebo respectively.
Time Frame: Baseline, Weeks 2,4,6,8,12,16,20,24
Population: "Number of participants analyzed": All randomized participants assigned to the study treatment. "Number analyzed" : Number of participants with observed data for each specified time point.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | PF-06651600 | PF-06700841 | Placebo
Number analyzed (Participants) | 48 | 47 | 47
units on a scale
  Week 2: number analyzed (Participants) | 48 | 47 | 46
  Week 2 | -0.74 [-2.06 to 0.59] | -0.93 [-2.27 to 0.40] | 1.18 [0.23 to 2.13]
  Week 4: number analyzed (Participants) | 48 | 47 | 44
  Week 4 | 2.93 [-1.32 to 7.17] | 7.70 [3.43 to 11.97] | 0.85 [-2.20 to 3.90]
  Week 6: number analyzed (Participants) | 47 | 45 | 43
  Week 6 | 12.44 [5.42 to 19.45] | 19.37 [12.29 to 26.45] | 1.32 [-3.72 to 6.35]
  Week 8: number analyzed (Participants) | 47 | 44 | 44
  Week 8 | 18.49 [9.57 to 27.41] | 29.30 [20.28 to 38.32] | 1.77 [-4.63 to 8.17]
  Week 12: number analyzed (Participants) | 47 | 44 | 45
  Week 12 | 24.49 [14.90 to 34.09] | 36.57 [26.86 to 46.29] | 1.62 [-5.26 to 8.50]
  Week 16: number analyzed (Participants) | 45 | 41 | 42
  Week 16 | 27.59 [17.67 to 37.50] | 41.16 [31.11 to 51.22] | 1.61 [-5.49 to 8.72]
  Week 20: number analyzed (Participants) | 45 | 40 | 40
  Week 20 | 29.32 [19.06 to 39.57] | 45.55 [35.14 to 55.97] | 1.62 [-5.73 to 8.98]
  Week 24: number analyzed (Participants) | 44 | 40 | 35
  Week 24 | 31.14 [20.79 to 41.49] | 49.18 [38.66 to 59.70] | 1.41 [-6.03 to 8.85]

9. Secondary Outcome: Percent Change From Baseline in Severity of Alopecia Tool (SALT) Across Time (Treatment Period)
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. The SALT score can vary from 0 to 100% with higher score indicates more severe disease. Baseline is defined as the last measurement prior to first dosing (Day 1). Percent change from baseline is defined as SALT baseline value minus SALT value at a specific visit divided by baseline and multiplying by 100. Positive change from baseline implies an improvement. Least Square Mean and 90% Confidence Interval of Arms (PF-06651600 and PF-06700841) are the Least Square Mean and 90% Confidence Interval for difference from placebo respectively.
Time Frame: Baseline, Weeks 2,4,6,8,12,16,20,24
Population: as for outcome 8
Measure: Least Squares Mean (90% Confidence Interval); unit: percent change
Arm/Group | PF-06651600 | PF-06700841 | Placebo
Number analyzed (Participants) | 48 | 47 | 47
percent change
  Week 2: number analyzed (Participants) | 48 | 47 | 46
  Week 2 | -0.76 [-2.26 to 0.75] | -1.13 [-2.64 to 0.39] | 1.26 [0.18 to 2.33]
  Week 4: number analyzed (Participants) | 48 | 47 | 44
  Week 4 | 3.99 [-0.86 to 8.83] | 9.70 [4.83 to 14.57] | 0.53 [-2.96 to 4.01]
  Week 6: number analyzed (Participants) | 47 | 45 | 43
  Week 6 | 15.88 [7.84 to 23.91] | 22.88 [14.77 to 30.99] | 1.02 [-4.75 to 6.80]
  Week 8: number analyzed (Participants) | 47 | 44 | 44
  Week 8 | 23.22 [13.15 to 33.29] | 34.78 [24.59 to 44.96] | 1.31 [-5.91 to 8.54]
  Week 12: number analyzed (Participants) | 47 | 44 | 45
  Week 12 | 30.99 [19.93 to 42.05] | 44.17 [32.97 to 55.37] | 0.99 [-6.94 to 8.92]
  Week 16: number analyzed (Participants) | 45 | 41 | 42
  Week 16 | 35.14 [23.65 to 46.62] | 49.99 [38.35 to 61.64] | 0.86 [-7.38 to 9.09]
  Week 20: number analyzed (Participants) | 45 | 40 | 40
  Week 20 | 37.31 [25.37 to 49.25] | 55.46 [43.34 to 67.58] | 0.91 [-7.65 to 9.47]
  Week 24: number analyzed (Participants) | 44 | 40 | 35
  Week 24 | 39.67 [27.66 to 51.68] | 59.71 [47.51 to 71.92] | 0.43 [-8.20 to 9.06]

10. Secondary Outcome: Percentage of Participants Achieving SALT 30 Across Time (Treatment Period)
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. A SALT 30 response is a 30% or greater reduction from baseline in SALT score. The SALT score can vary from 0 to 100%, with higher scores representing increasing severity of disease. The analysis was done using FAS (full analysis set) based on Non-responder imputation (ie. set missing values to be non-responsive) data. The percentage(Number) and 90% confidence interval (CI) of Arms(PF-06651600 and PF-06700841) in this outcome measurement is the percentage and 90% CI for difference from placebo. The 90% CI was calculated using Chan and Zhang method.
Time Frame: Baseline, Weeks 2,4,6,8,12,16,20,24
Population: All participants in the Full analysis set (FAS) was used. FAS consisted of all randomized participants, assigned to the randomized treatment regardless of what treatment, if any, was received.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06651600 | PF-06700841 | Placebo
Number analyzed (Participants) | 48 | 47 | 47
percentage of participants
  Week 2 | -2.1 [-9.7 to 3.7] | -2.1 [-9.7 to 3.5] | 2.1 [0.2 to 8.8]
  Week 4 | 6.2 [-2.3 to 15.8] | 12.8 [3.0 to 24.0] | 2.1 [0.2 to 8.8]
  Week 6 | 18.7 [7.0 to 31.0] | 27.7 [15.4 to 40.4] | 2.1 [0.2 to 8.8]
  Week 8 | 25.0 [13.2 to 37.4] | 38.3 [25.8 to 51.4] | 2.1 [0.2 to 8.8]
  Week 12 | 39.5 [26.4 to 52.6] | 48.9 [35.8 to 61.8] | 2.1 [0.2 to 8.8]
  Week 16 | 45.8 [32.2 to 58.7] | 55.3 [42.0 to 67.8] | 2.1 [0.2 to 8.8]
  Week 20 | 47.9 [34.2 to 60.7] | 59.6 [46.3 to 71.7] | 2.1 [0.2 to 8.8]
  Week 24 | 47.9 [34.2 to 60.7] | 61.7 [48.2 to 73.6] | 2.1 [0.2 to 8.8]

11. Secondary Outcome: Percentage of Participants Achieving SALT 50 Across Time (Treatment Period)
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. A SALT 50 response is a 50% or greater reduction from baseline in SALT score. The SALT score can vary from 0 to 100%, with higher scores representing increasing severity of disease. The analysis was done using FAS (full analysis set) based on Non-responder imputation (ie. set missing values to be non-responsive) data. The percentage(Number) and 90% confidence interval (CI) of Arms(PF-06651600 and PF-06700841) in this outcome measurement is the percentage and 90% CI for difference from placebo. The 90% CI was calculated using Chan and Zhang method.
Time Frame: Baseline, Weeks 2,4,6,8,12,16,20,24
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06651600 | PF-06700841 | Placebo
Number analyzed (Participants) | 48 | 47 | 47
percentage of participants
  Week 2 | 0.0 [-6.2 to 6.1] | 0.0 [-6.2 to 6.2] | 0 [0.0 to 5.7]
  Week 4 | 0.0 [-6.2 to 6.1] | 10.6 [3.6 to 21.1] | 0 [0.0 to 5.7]
  Week 6 | 10.4 [1.1 to 21.1] | 17.0 [6.5 to 28.8] | 2.1 [0.2 to 8.8]
  Week 8 | 18.7 [7.0 to 31.0] | 29.8 [17.2 to 42.7] | 2.1 [0.2 to 8.8]
  Week 12 | 27.0 [15.0 to 39.6] | 36.2 [23.8 to 49.2] | 2.1 [0.2 to 8.8]
  Week 16 | 33.3 [20.3 to 46.2] | 40.4 [27.8 to 53.5] | 2.1 [0.2 to 8.8]
  Week 20 | 33.3 [20.3 to 46.2] | 46.8 [33.8 to 59.8] | 2.1 [0.2 to 8.8]
  Week 24 | 37.5 [24.5 to 50.6] | 51.1 [37.9 to 63.8] | 2.1 [0.2 to 8.8]

12. Secondary Outcome: Percentage of Participants Achieving SALT 75 Across Time (Treatment Period)
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. A SALT 75 response is a 75% or greater reduction from baseline in SALT score. The SALT score can vary from 0 to 100%, with higher scores representing increasing severity of disease. The analysis was done using FAS (full analysis set) based on Non-responder imputation (ie. set missing values to be non-responsive) data. The percentage(Number) and 90% confidence interval (CI) of Arms(PF-06651600 and PF-06700841) in this outcome measurement is the percentage and 90% CI for difference from placebo. The 90% CI was calculated using Chan and Zhang method.
Time Frame: Baseline, Weeks 2,4,6,8,12,16,20,24
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06651600 | PF-06700841 | Placebo
Number analyzed (Participants) | 48 | 47 | 47
percentage of participants
  Week 2 | 0.0 [-6.2 to 6.1] | 0.0 [-6.2 to 6.2] | 0 [0.0 to 5.7]
  Week 4 | 0.0 [-6.2 to 6.1] | 0.0 [-6.2 to 6.2] | 0 [0.0 to 5.7]
  Week 6 | 8.3 [1.8 to 18.1] | 10.6 [3.6 to 21.1] | 0 [0.0 to 5.7]
  Week 8 | 12.5 [2.8 to 23.6] | 23.4 [11.8 to 36.2] | 2.1 [0.2 to 8.8]
  Week 12 | 16.6 [6.3 to 28.6] | 27.7 [15.4 to 40.4] | 2.1 [0.2 to 8.8]
  Week 16 | 20.8 [8.6 to 33.0] | 31.9 [19.0 to 44.9] | 2.1 [0.2 to 8.8]
  Week 20 | 25.0 [13.2 to 37.4] | 38.3 [25.8 to 51.4] | 2.1 [0.2 to 8.8]
  Week 24 | 27.0 [15.0 to 39.6] | 40.4 [27.8 to 53.5] | 2.1 [0.2 to 8.8]

13. Secondary Outcome: Percentage of Participants Achieving SALT 90 Across Time (Treatment Period)
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. A SALT 90 response is a 90% or greater reduction from baseline in SALT score. The SALT score can vary from 0 to 100%, with higher scores representing increasing severity of disease. The analysis was done using FAS (full analysis set) based on Non-responder imputation (ie. set missing values to be non-responsive) data. The percentage(Number) and 90% confidence interval (CI) of Arms(PF-06651600 and PF-06700841) in this outcome measurement is the percentage and 90% CI for difference from placebo. The 90% CI was calculated using Chan and Zhang method.
Time Frame: Baseline, Weeks 2,4,6,8,12,16,20,24
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06651600 | PF-06700841 | Placebo
Number analyzed (Participants) | 48 | 47 | 47
percentage of participants
  Week 2 | 0.0 [-6.2 to 6.1] | 0.0 [-6.2 to 6.2] | 0 [0.0 to 5.7]
  Week 4 | 0.0 [-6.2 to 6.1] | 0.0 [-6.2 to 6.2] | 0 [0.0 to 5.7]
  Week 6 | 0.0 [-6.2 to 6.1] | 6.4 [0.2 to 15.7] | 0 [0.0 to 5.7]
  Week 8 | 4.2 [-2.0 to 12.5] | 12.8 [5.2 to 23.6] | 0 [0.0 to 5.7]
  Week 12 | 10.4 [3.4 to 20.7] | 25.5 [15.4 to 38.1] | 0 [0.0 to 5.7]
  Week 16 | 16.7 [8.6 to 27.7] | 27.7 [17.2 to 40.3] | 0 [0.0 to 5.7]
  Week 20 | 18.7 [7.0 to 31.0] | 29.8 [17.2 to 42.7] | 2.1 [0.2 to 8.8]
  Week 24 | 25.0 [15.1 to 37.3] | 34.0 [22.7 to 47.0] | 0 [0.0 to 5.7]

14. Secondary Outcome: Percentage of Participants Achieving SALT 100 Across Time (Treatment Period)
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. A SALT 100 response is a 100% or greater reduction from baseline in SALT score. The SALT score can vary from 0 to 100%, with higher scores representing increasing severity of disease. The analysis was done using FAS (full analysis set) based on Non-responder imputation (ie. set missing values to be non-responsive) data. The percentage(Number) and 90% confidence interval (CI) of Arms(PF-06651600 and PF-06700841) in this outcome measurement is the percentage and 90% CI for difference from placebo. The 90% CI was calculated using Chan and Zhang method.
Time Frame: Baseline, Weeks 2,4,6,8,12,16,20,24
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | PF-06651600 | PF-06700841 | Placebo
Number analyzed (Participants) | 48 | 47 | 47
percentage of participants
  Week 2 | 0.0 [-6.2 to 6.1] | 0.0 [-6.2 to 6.2] | 0 [0.0 to 5.7]
  Week 4 | 0.0 [-6.2 to 6.1] | 0.0 [-6.2 to 6.2] | 0 [0.0 to 5.7]
  Week 6 | 0.0 [-6.2 to 6.1] | 0.0 [-6.2 to 6.2] | 0 [0.0 to 5.7]
  Week 8 | 0.0 [-6.2 to 6.1] | 2.1 [-3.5 to 9.7] | 0 [0.0 to 5.7]
  Week 12 | 2.1 [-3.8 to 9.5] | 6.4 [0.2 to 15.7] | 0 [0.0 to 5.7]
  Week 16 | 2.1 [-3.8 to 9.5] | 8.5 [1.9 to 18.4] | 0 [0.0 to 5.7]
  Week 20 | 4.2 [-2.0 to 12.5] | 12.8 [5.2 to 23.6] | 0 [0.0 to 5.7]
  Week 24 | 12.5 [5.1 to 23.2] | 12.8 [5.2 to 23.6] | 0 [0.0 to 5.7]

15. Secondary Outcome: Number of Participants With the IGA Score Change (Treatment Period)
Description: The clinical evaluator of alopecia areata (AA) will perform an assessment of the overall improvement of AA and assign an Investigator Global Assessment (IGA) score(ranging from 0 to 5) with higher score representing higher regrowth rate. Baseline is defined as the last measurement prior to first dosing (Day 1).
Time Frame: baseline, Week 2,4,6,8,12,16,20,24
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 | PF-06700841 | Placebo
Number analyzed (Participants) | 48 | 47 | 47
Participants
  Baseline: 0 (NO CHANGE OR FURTHER LOSS) | 48 | 47 | 47
  Baseline: 1 (1-24% REGROWTH) | 0 | 0 | 0
  Baseline: 2 (25-49% REGROWTH) | 0 | 0 | 0
  Baseline: 3 (50-74% REGROWTH) | 0 | 0 | 0
  Baseline: 4 (75-99% REGROWTH) | 0 | 0 | 0
  Baseline: 5 (100% REGROWTH) | 0 | 0 | 0
  Week 2: number analyzed (Participants) | 48 | 47 | 46
  Week 2: 0 (NO CHANGE OR FURTHER LOSS) | 40 | 43 | 40
  Week 2: 1 (1-24% REGROWTH) | 8 | 4 | 5
  Week 2: 2 (25-49% REGROWTH) | 0 | 0 | 1
  Week 2: 3 (50-74% REGROWTH) | 0 | 0 | 0
  Week 2: 4 (75-99% REGROWTH) | 0 | 0 | 0
  Week 2: 5 (100% REGROWTH) | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 48 | 47 | 43
  Week 4: 0 (NO CHANGE OR FURTHER LOSS) | 29 | 21 | 36
  Week 4: 1 (1-24% REGROWTH) | 15 | 19 | 6
  Week 4: 2 (25-49% REGROWTH) | 4 | 2 | 1
  Week 4: 3 (50-74% REGROWTH) | 0 | 5 | 0
  Week 4: 4 (75-99% REGROWTH) | 0 | 0 | 0
  Week 4: 5 (100% REGROWTH) | 0 | 0 | 0
  Week 6: number analyzed (Participants) | 47 | 45 | 43
  Week 6: 0 (NO CHANGE OR FURTHER LOSS) | 16 | 10 | 35
  Week 6: 1 (1-24% REGROWTH) | 18 | 17 | 6
  Week 6: 2 (25-49% REGROWTH) | 7 | 9 | 1
  Week 6: 3 (50-74% REGROWTH) | 2 | 4 | 1
  Week 6: 4 (75-99% REGROWTH) | 4 | 5 | 0
  Week 6: 5 (100% REGROWTH) | 0 | 0 | 0
  Week 8: number analyzed (Participants) | 47 | 44 | 44
  Week 8: 0 (NO CHANGE OR FURTHER LOSS) | 13 | 7 | 33
  Week 8: 1 (1-24% REGROWTH) | 17 | 17 | 9
  Week 8: 2 (25-49% REGROWTH) | 7 | 5 | 1
  Week 8: 3 (50-74% REGROWTH) | 3 | 3 | 0
  Week 8: 4 (75-99% REGROWTH) | 7 | 11 | 1
  Week 8: 5 (100% REGROWTH) | 0 | 1 | 0
  Week 12: number analyzed (Participants) | 47 | 44 | 45
  Week 12: 0 (NO CHANGE OR FURTHER LOSS) | 13 | 6 | 33
  Week 12: 1 (1-24% REGROWTH) | 11 | 11 | 10
  Week 12: 2 (25-49% REGROWTH) | 9 | 9 | 1
  Week 12: 3 (50-74% REGROWTH) | 5 | 4 | 0
  Week 12: 4 (75-99% REGROWTH) | 8 | 10 | 1
  Week 12: 5 (100% REGROWTH) | 1 | 4 | 0
  Week 16: number analyzed (Participants) | 45 | 41 | 42
  Week 16: 0 (NO CHANGE OR FURTHER LOSS) | 14 | 5 | 31
  Week 16: 1 (1-24% REGROWTH) | 7 | 7 | 9
  Week 16: 2 (25-49% REGROWTH) | 7 | 9 | 1
  Week 16: 3 (50-74% REGROWTH) | 6 | 4 | 0
  Week 16: 4 (75-99% REGROWTH) | 10 | 11 | 1
  Week 16: 5 (100% REGROWTH) | 1 | 5 | 0
  Week 20: number analyzed (Participants) | 45 | 40 | 40
  Week 20: 0 (NO CHANGE OR FURTHER LOSS) | 14 | 4 | 29
  Week 20: 1 (1-24% REGROWTH) | 6 | 6 | 9
  Week 20: 2 (25-49% REGROWTH) | 8 | 7 | 1
  Week 20: 3 (50-74% REGROWTH) | 4 | 4 | 0
  Week 20: 4 (75-99% REGROWTH) | 10 | 11 | 1
  Week 20: 5 (100% REGROWTH) | 3 | 8 | 0
  Week 24: number analyzed (Participants) | 44 | 40 | 35
  Week 24: 0 (NO CHANGE OR FURTHER LOSS) | 13 | 4 | 27
  Week 24: 1 (1-24% REGROWTH) | 5 | 6 | 6
  Week 24: 2 (25-49% REGROWTH) | 7 | 5 | 1
  Week 24: 3 (50-74% REGROWTH) | 5 | 5 | 0
  Week 24: 4 (75-99% REGROWTH) | 8 | 13 | 1
  Week 24: 5 (100% REGROWTH) | 6 | 7 | 0

16. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (All-causality and Treatment-related) - Treatment Period
Description: as for outcome 4
Time Frame: baseline up to Week 24
Population: All participants who received at least 1 dose of investigational product (PF-06651600, PF-06700841 or placebo) in Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 | PF-06700841 | Placebo
Number analyzed (Participants) | 48 | 47 | 47
Participants
  TEAE (All Causalities) | 32 | 36 | 35
  TEAE (Treatment Related) | 13 | 20 | 14

17. Secondary Outcome: Number of Participants With Laboratory Abnormalities During Treatment Period
Description: as for outcome 5
Time Frame: Baseline up to Week 24
Population: All participants in safety analysis set (SAS) who received at least 1 dose of investigational product (PF-06651600, PF-06700841 or placebo) and had abnormal laboratory data in treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06651600 | PF-06700841 | Placebo
Number analyzed (Participants) | 48 | 47 | 46
Participants
  With abnormalities without regard to baseline | 35 | 36 | 32
  Meeting Safety Criteria | 12 | 29 | 5
  Meeting Retest Criteria | 5 | 18 | 9
  Meeting Discontinuation Criteria | 0 | 3 | 0

18. Secondary Outcome: Time to Achieve the Retreatment Criteria During the Withdrawal/Retreatment Part of the Extension Period Among Subjects Who Achieved Primary Endpoint at Week 24 (SBE Period)
Description: Time to re-treatment (weeks) = (date of re-treatment criteria met - date at Week 24 +1)/7. The calendar time to retreatment was calculated. Baseline is defined as Week 24 measurement. The duration in Drug Holiday #1 (ranging from 2-6 weeks) is counted in the Kaplan-Meier analysis. One subject directly entered the re-treatment period and hence is censored at baseline in the Kaplan-Meier analysis.
Time Frame: Week 24 up to Week 52
Population: All randomized participants who were responsive at Week 24 (ie, achieving SALT30 at Week 24).All randomized participants who were responsive at Week 24 (ie, achieving SALT30 at Week 24).
Measure: Number (95% Confidence Interval); unit: Weeks
Groups:
- PF-06651600 Responders: Participants received PF-06651600 200 mg once daily (QD) for 4 weeks induction period followed by PF-06651600 50 mg QD for a 20 weeks maintenance period responsive at Week 24 (ie, achieving SALT 30) who were assigned to placebo (withdrawal)
- PF-06700841 Responders: Participants received PF-06700841 60 mg tablets QD for a 4-week induction period followed by PF-06700841 30 mg tablets QD for a 20-week maintenance period and responsive at Week 24 (ie, achieving SALT 30) who were assigned to placebo (withdrawal)
Arm/Group | PF-06651600 Responders | PF-06700841 Responders
Number analyzed (Participants) | 22 | 24
Weeks
  Q1 time to retreatment (25th percentile of time) | 10.1 [4.3 to 12.6] | 11.0 [4.1 to 16.1]
  Median time to retreatment | 16.1 [10.1 to 20.3] | 24.1 [14.6 to NA] — NA indicates not estimable. The withdrawal segment is not lengthy enough to observe upper limit of the 95% CI for the median time to retreatment (ie. 50% of participants meeting the criterion).
  Q3 time to retreatment (75th percentile of time) | 21.1 [16.1 to NA] — NA indicates not estimable. The withdrawal segment is not lengthy enough to observe upper limit of the 95% CI for the Q3 time to retreatment (ie. 75% of participants meeting the criterion). | NA [24.3 to NA] — NA indicates not estimable. The withdrawal segment is not lengthy enough to observe Q3 time to retreatment (ie. 75% of participants meeting the criterion) and corresponding upper limit of the 95% CI.

19. Secondary Outcome: Change From Baseline in SALT Across Time (SBE Period)
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. The SALT score can vary from 0 to 100% with higher score indicates more severe disease. Baseline is defined as the last measurement prior to first dosing (Day 1). Change from baseline is defined as the baseline value minus the value at a specific visit. Positive change from baseline implies an improvement. Least Square Mean and 90% confidence interval in this outcome measurement is the LSM and 90%CI for difference from initial 24-week treatment period placebo respectively.
Time Frame: Weeks 30, 32, 34, 36, 40, 44, 48, 52 for non-responders, and AT Weeks 2, 4, 6, 8, 12, 16, 20, 24 for retreated responders.(AT=active treatment)
Population: Number of Participants Analyzed: All randomized participants assigned to the study treatment. Number Analyzed: Number of Participants with observed data. 6 groups of participants were each compared with initial 24-week treatment period placebo.
Measure: Least Squares Mean (90% Confidence Interval); unit: unit on a scale
Arm/Group | Active Non-responders on PF-06651600 | Active Non-responders on PF-06700841 | Placebo Non-responders on PF-06651600 | Placebo Non-responders on PF-06700841 | Retreated PF-06651600 Responders in the Retreatment Segment | Retreated Responders on PF-06700841 in the Retreatment Segment
Number analyzed (Participants) | 16 | 5 | 17 | 12 | 14 | 15
unit on a scale
  Week 30/ AT Week 2: number analyzed (Participants) | 15 | 5 | 16 | 10 | 13 | 14
  Week 30/ AT Week 2 | 1.76 [-4.47 to 7.99] | 0.09 [-9.83 to 10.01] | 2.99 [-4.56 to 10.54] | -0.31 [-9.53 to 8.92] | 25.04 [15.01 to 35.08] | 19.83 [10.00 to 29.66]
  Week 32/ AT Week 4: number analyzed (Participants) | 16 | 4 | 17 | 12 | 14 | 14
  Week 32/ AT Week 4 | 1.85 [-4.37 to 8.07] | 2.22 [-7.78 to 12.21] | 3.37 [-4.06 to 10.79] | 3.71 [-4.93 to 12.35] | 27.63 [17.67 to 37.59] | 15.66 [5.82 to 25.51]
  Week 34/ AT Week 6: number analyzed (Participants) | 16 | 4 | 16 | 12 | 13 | 13
  Week 34/ AT Week 6 | 1.80 [-4.42 to 8.02] | 3.16 [-6.90 to 13.23] | 10.16 [2.55 to 17.77] | 24.67 [16.00 to 33.34] | 33.78 [23.72 to 43.83] | 20.09 [10.17 to 30.02]
  Week 36/ AT Week 8: number analyzed (Participants) | 14 | 4 | 16 | 11 | 13 | 13
  Week 36/ AT Week 8 | 2.16 [-4.09 to 8.40] | 3.01 [-7.12 to 13.14] | 8.93 [1.34 to 16.52] | 42.32 [33.37 to 51.28] | 38.80 [28.75 to 48.84] | 27.35 [17.42 to 37.27]
  Week 40/ AT Week 12: number analyzed (Participants) | 13 | 4 | 16 | 12 | 12 | 13
  Week 40/ AT Week 12 | 3.35 [-2.91 to 9.61] | 3.19 [-7.00 to 13.38] | 18.30 [10.73 to 25.86] | 50.27 [41.65 to 58.90] | 43.70 [33.58 to 53.82] | 39.28 [29.36 to 49.19]
  Week 44/ AT Week 16: number analyzed (Participants) | 15 | 3 | 14 | 11 | 10 | 11
  Week 44/ AT Week 16 | 3.41 [-2.84 to 9.67] | 3.12 [-7.19 to 13.43] | 25.71 [17.70 to 33.72] | 54.69 [45.73 to 63.64] | 48.93 [38.59 to 59.27] | 50.58 [40.48 to 60.69]
  Week 48/ AT Week 20: number analyzed (Participants) | 15 | 3 | 15 | 10 | 10 | 10
  Week 48/ AT Week 20 | 4.70 [-1.57 to 10.97] | 2.97 [-7.39 to 13.34] | 25.28 [17.42 to 33.13] | 62.45 [53.13 to 71.77] | 53.74 [43.39 to 64.09] | 53.79 [43.57 to 64.02]
  Week 52/ AT Week 24: number analyzed (Participants) | 13 | 3 | 12 | 11 | 9 | 10
  Week 52/ AT Week 24 | 7.06 [0.75 to 13.38] | 3.01 [-7.47 to 13.49] | 28.88 [20.20 to 37.56] | 58.53 [49.42 to 67.63] | 55.94 [45.42 to 66.46] | 58.37 [48.11 to 68.64]

20. Secondary Outcome: Percentage of Participants Achieving SALT 30 Across Time (SBE Period)
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. A SALT 30 response is a 30% or greater reduction from baseline in SALT score. The SALT score can vary from 0 to 100%, with higher scores representing increasing severity of disease. The analysis was done using FAS (full analysis set) based on Non-responder imputation (ie. set missing values to be non-responsive) data. The percentage(Number) and 90% confidence interval (CI) in this outcome measurement is the percentage and 90% CI for difference from initial 24-week treatment period placebo. The 90% CI was calculated using Chan and Zhang method.
Time Frame: as for outcome 19
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: percent of participants
Arm/Group | Active Non-responders on PF-06651600 | Active Non-responders on PF-06700841 | Placebo Non-responders on PF-06651600 | Placebo Non-responders on PF-06700841 | Retreated PF-06651600 Responders in the Retreatment Segment | Retreated Responders on PF-06700841 in the Retreatment Segment
Number analyzed (Participants) | 16 | 5 | 17 | 12 | 14 | 15
percent of participants
  Week 30/ AT Week 2 | 4.1 [-5.3 to 23.0] | -2.1 [-10.9 to 40.0] | 3.8 [-5.5 to 21.6] | -2.1 [-9.7 to 18.9] | 47.9 [25.3 to 70.0] | 31.2 [12.8 to 54.0]
  Week 32/ AT Week 4 | 4.1 [-5.3 to 23.0] | -2.1 [-10.9 to 40.0] | 9.6 [-2.4 to 30.2] | 14.5 [0.4 to 39.4] | 62.2 [38.2 to 81.5] | 11.2 [-1.0 to 33.5]
  Week 34/ AT Week 6 | 4.1 [-5.3 to 23.0] | -2.1 [-10.9 to 40.0] | 21.4 [4.8 to 43.2] | 31.2 [10.9 to 57.0] | 69.3 [45.3 to 86.5] | 31.2 [12.8 to 54.0]
  Week 36/ AT Week 8 | 4.1 [-5.3 to 23.0] | -2.1 [-10.9 to 40.0] | 21.4 [4.8 to 43.2] | 56.2 [30.8 to 78.2] | 69.3 [45.3 to 86.5] | 44.5 [23.2 to 66.5]
  Week 40/ AT Week 12 | 10.4 [-1.5 to 31.8] | -2.1 [-10.9 to 40.0] | 27.3 [8.5 to 49.6] | 81.2 [55.6 to 94.4] | 62.2 [38.2 to 81.5] | 51.2 [28.9 to 72.2]
  Week 44/ AT Week 16 | 10.4 [-1.5 to 31.8] | -2.1 [-10.9 to 40.0] | 33.2 [15.2 to 54.5] | 64.5 [38.4 to 84.5] | 62.2 [38.2 to 81.5] | 51.2 [28.9 to 72.2]
  Week 48/ AT Week 20 | 10.4 [-1.5 to 31.8] | -2.1 [-10.9 to 40.0] | 39.0 [20.0 to 60.1] | 64.5 [38.4 to 84.5] | 69.3 [45.3 to 86.5] | 51.2 [28.9 to 72.2]
  Week 52/ AT Week 24 | 10.4 [-1.5 to 31.8] | -2.1 [-10.9 to 40.0] | 27.3 [8.5 to 49.6] | 64.5 [38.4 to 84.5] | 55.0 [31.6 to 76.0] | 51.2 [28.9 to 72.2]

21. Secondary Outcome: Percentage of Participants Achieving SALT 50 Across Time (SBE Period)
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. A SALT 50 response is a 50% or greater reduction from baseline in SALT score. The SALT score can vary from 0 to 100%, with higher scores representing increasing severity of disease. The analysis was done using FAS (full analysis set) based on Non-responder imputation (ie. set missing values to be non-responsive) data. The percentage(Number) and 90% confidence interval (CI) in this outcome measurement is the percentage and 90% CI for difference from initial 24-week treatment period placebo. The 90% CI was calculated using Chan and Zhang method.
Time Frame: as for outcome 19
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Active Non-responders on PF-06651600 | Active Non-responders on PF-06700841 | Placebo Non-responders on PF-06651600 | Placebo Non-responders on PF-06700841 | Retreated PF-06651600 Responders in the Retreatment Segment | Retreated Responders on PF-06700841 in the Retreatment Segment
Number analyzed (Participants) | 16 | 5 | 17 | 12 | 14 | 15
percentage of participants
  Week 30/ AT Week 2 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 0.0 [-6.3 to 22.1] | 14.3 [2.4 to 38.5] | 20.0 [5.7 to 44.0]
  Week 32/ AT Week 4 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 0.0 [-6.3 to 22.1] | 21.4 [6.1 to 46.6] | 6.7 [-2.1 to 27.9]
  Week 34/ AT Week 6 | -2.1 [-9.7 to 13.8] | -2.1 [-10.9 to 40.0] | 9.6 [-2.4 to 30.2] | 31.2 [10.9 to 57.0] | 26.4 [6.1 to 50.0] | 11.2 [-1.0 to 33.5]
  Week 36/ AT Week 8 | -2.1 [-9.7 to 13.8] | -2.1 [-10.9 to 40.0] | 3.8 [-5.5 to 21.6] | 56.2 [30.8 to 78.2] | 33.6 [14.1 to 57.2] | 24.5 [5.6 to 47.1]
  Week 40/ AT Week 12 | -2.1 [-9.7 to 13.8] | -2.1 [-10.9 to 40.0] | 15.5 [1.1 to 36.8] | 56.2 [30.8 to 78.2] | 47.9 [25.3 to 70.0] | 44.5 [23.2 to 66.5]
  Week 44/ AT Week 16 | -2.1 [-9.7 to 13.8] | -2.1 [-10.9 to 40.0] | 21.4 [4.8 to 43.2] | 64.5 [38.4 to 84.5] | 47.9 [25.3 to 70.0] | 44.5 [23.2 to 66.5]
  Week 48/ AT Week 20 | 4.1 [-5.3 to 23.0] | -2.1 [-10.9 to 40.0] | 27.3 [8.5 to 49.6] | 64.5 [38.4 to 84.5] | 47.9 [25.3 to 70.0] | 37.9 [17.9 to 60.3]
  Week 52/ AT Week 24 | 4.1 [-5.3 to 23.0] | -2.1 [-10.9 to 40.0] | 27.3 [8.5 to 49.6] | 64.5 [38.4 to 84.5] | 47.9 [25.3 to 70.0] | 44.5 [23.2 to 66.5]

22. Secondary Outcome: Percentage of Participants Achieving SALT 75 Across Time (SBE Period)
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. A SALT 75 response is a 75% or greater reduction from baseline in SALT score. The SALT score can vary from 0 to 100%, with higher scores representing increasing severity of disease. The analysis was done using FAS (full analysis set) based on Non-responder imputation (ie. set missing values to be non-responsive) data. The percentage(Number) and 90% confidence interval (CI) in this outcome measurement is the percentage and 90% CI for difference from initial 24-week treatment period placebo. The 90% CI was calculated using Chan and Zhang method.
Time Frame: as for outcome 19
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Active Non-responders on PF-06651600 | Active Non-responders on PF-06700841 | Placebo Non-responders on PF-06651600 | Placebo Non-responders on PF-06700841 | Retreated PF-06651600 Responders in the Retreatment Segment | Retreated Responders on PF-06700841 in the Retreatment Segment
Number analyzed (Participants) | 16 | 5 | 17 | 12 | 14 | 15
percentage of participants
  Week 30/ AT Week 2 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 0.0 [-6.3 to 22.1] | 0.0 [-6.8 to 19.3] | 0.0 [-6.6 to 18.1]
  Week 32/ AT Week 4 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 0.0 [-6.3 to 22.1] | 7.1 [-1.9 to 29.7] | 0.0 [-6.6 to 18.1]
  Week 34/ AT Week 6 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 8.3 [-1.5 to 33.9] | 14.3 [2.4 to 38.5] | 6.7 [-2.1 to 27.9]
  Week 36/ AT Week 8 | -2.1 [-9.7 to 13.8] | -2.1 [-10.9 to 40.0] | -2.1 [-9.7 to 13.3] | 22.9 [2.8 to 48.7] | 26.4 [6.1 to 50.0] | 17.9 [1.8 to 40.6]
  Week 40/ AT Week 12 | -2.1 [-9.7 to 13.8] | -2.1 [-10.9 to 40.0] | 3.8 [-5.5 to 21.6] | 39.5 [17.0 to 64.5] | 26.4 [6.1 to 50.0] | 31.2 [12.8 to 54.0]
  Week 44/ AT Week 16 | -2.1 [-9.7 to 13.8] | -2.1 [-10.9 to 40.0] | 15.5 [1.1 to 36.8] | 56.2 [30.8 to 78.2] | 26.4 [6.1 to 50.0] | 37.9 [17.9 to 60.3]
  Week 48/ AT Week 20 | -2.1 [-9.7 to 13.8] | -2.1 [-10.9 to 40.0] | 15.5 [1.1 to 36.8] | 64.5 [38.4 to 84.5] | 28.6 [6.1 to 50.0] | 37.9 [17.9 to 60.3]
  Week 52/ AT Week 24 | 4.1 [-5.3 to 23.0] | -2.1 [-10.9 to 40.0] | 27.3 [8.5 to 49.6] | 64.5 [38.4 to 84.5] | 33.6 [14.1 to 57.2] | 37.9 [17.9 to 60.3]

23. Secondary Outcome: Percentage of Participants Achieving SALT 90 Across Time (SBE Period)
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. A SALT 90 response is a 90% or greater reduction from baseline in SALT score. The SALT score can vary from 0 to 100%, with higher scores representing increasing severity of disease. The analysis was done using FAS (full analysis set) based on Non-responder imputation (ie. set missing values to be non-responsive) data. The percentage(Number) and 90% confidence interval (CI) in this outcome measurement is the percentage and 90% CI for difference from initial 24-week treatment period placebo. The 90% CI was calculated using Chan and Zhang method.
Time Frame: as for outcome 19
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Active Non-responders on PF-06651600 | Active Non-responders on PF-06700841 | Placebo Non-responders on PF-06651600 | Placebo Non-responders on PF-06700841 | Retreated PF-06651600 Responders in the Retreatment Segment | Retreated Responders on PF-06700841 in the Retreatment Segment
Number analyzed (Participants) | 16 | 5 | 17 | 12 | 14 | 15
percentage of participants
  Week 30/ AT Week 2 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 0.0 [-6.3 to 22.1] | 0.0 [-6.8 to 19.3] | 0.0 [-6.6 to 18.1]
  Week 32/ AT Week 4 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 0.0 [-6.3 to 22.1] | 0.0 [-6.8 to 19.3] | 0.0 [-6.6 to 18.1]
  Week 34/ AT Week 6 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 0.0 [-6.3 to 22.1] | 0.0 [-6.8 to 19.3] | 0.0 [-6.6 to 18.1]
  Week 36/ AT Week 8 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 8.3 [-1.5 to 33.9] | 7.1 [-1.9 to 29.7] | 6.7 [-2.1 to 27.9]
  Week 40/ AT Week 12 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 25.0 [7.2 to 52.7] | 14.3 [2.4 to 38.5] | 13.3 [2.1 to 36.3]
  Week 44/ AT Week 16 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 33.3 [12.3 to 60.9] | 21.4 [6.1 to 46.6] | 20.0 [5.7 to 44.0]
  Week 48/ AT Week 20 | -2.1 [-9.7 to 13.8] | -2.1 [-10.9 to 40.0] | 3.8 [-5.5 to 21.6] | 47.9 [23.6 to 71.6] | 26.4 [6.1 to 50.0] | 24.5 [5.6 to 47.1]
  Week 52/ AT Week 24 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 17.6 [5.0 to 39.6] | 50.0 [24.5 to 75.5] | 28.6 [10.4 to 54.0] | 40.0 [19.1 to 64.0]

24. Secondary Outcome: Percentage of Participants Achieving SALT 100 Across Time (SBE Period)
Description: SALT is a quantitative assessment of alopecia areata (AA) severity based on the scalp hair loss. A SALT 100 response is a 100% or greater reduction from baseline in SALT score. The SALT score can vary from 0 to 100%, with higher scores representing increasing severity of disease. The analysis was done using FAS (full analysis set) based on Non-responder imputation (ie. set missing values to be non-responsive) data. The percentage(Number) and 90% confidence interval (CI) in this outcome measurement is the percentage and 90% CI for difference from initial 24-week treatment period placebo. The 90% CI was calculated using Chan and Zhang method.
Time Frame: as for outcome 19
Population: as for outcome 10
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Active Non-responders on PF-06651600 | Active Non-responders on PF-06700841 | Placebo Non-responders on PF-06651600 | Placebo Non-responders on PF-06700841 | Retreated PF-06651600 Responders in the Retreatment Segment | Retreated Responders on PF-06700841 in the Retreatment Segment
Number analyzed (Participants) | 16 | 5 | 17 | 12 | 14 | 15
percentage of participants
  Week 30/ AT Week 2 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 0.0 [-6.3 to 22.1] | 0.0 [-6.8 to 19.3] | 0.0 [-6.6 to 18.1]
  Week 32/ AT Week 4 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 0.0 [-6.3 to 22.1] | 0.0 [-6.8 to 19.3] | 0.0 [-6.6 to 18.1]
  Week 34/ AT Week 6 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 0.0 [-6.3 to 22.1] | 0.0 [-6.8 to 19.3] | 0.0 [-6.6 to 18.1]
  Week 36/ AT Week 8 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 0.0 [-6.3 to 22.1] | 0.0 [-6.8 to 19.3] | 0.0 [-6.6 to 18.1]
  Week 40/ AT Week 12 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 8.3 [-1.5 to 33.9] | 7.1 [-1.9 to 29.7] | 0.0 [-6.6 to 18.1]
  Week 44/ AT Week 16 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 8.3 [-1.5 to 33.9] | 7.1 [-1.9 to 29.7] | 13.3 [2.1 to 36.3]
  Week 48/ AT Week 20 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 8.3 [-1.5 to 33.9] | 7.1 [-1.9 to 29.7] | 20.0 [5.7 to 44.0]
  Week 52/ AT Week 24 | 0.0 [-6.3 to 17.1] | 0.0 [-7.4 to 45.1] | 0.0 [-6.2 to 16.2] | 8.3 [-1.5 to 33.9] | 14.3 [2.4 to 38.5] | 20.0 [5.7 to 44.0]

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 113 weeks
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study.
  Participants were counted only once per treatment per event.
Groups:
- Treatment Period-Placebo: Participants received placebo tablets QD both matching for PF-06651600 and PF-06700841
- Treatment Period-PF-06651600: Participants received PF-06651600 200 mg tablets QD for a 4-week induction period followed by PF-06651600 50 mg tablets QD for a 20-week maintenance period.
- Treatment Period-PF-06700841: Participants received PF-06700841 60 mg tablets QD for a 4-week induction period followed by PF-06700841 30 mg tablets QD for a 20-week maintenance period.
- Single Blind Extension-Active Non-responders on PF-06651600: Participants initially treated with PF-06651600 in the Initial 24-Week Treatment Period and not responsive at Week 24 (ie, not achieving ≥30% improvement from baseline in SALT [SALT 30]) who were continually assigned to PF-06651600 in the Non-Responder Segment of the SBE Period
- Single Blind Extension-Placebo Non-responders on PF-06651600: Participants initially treated with placebo in the Initial 24-Week Treatment Period (1 participant receiving placebo in the Initial 24-Week Treatment Period was responsive at Week 24 but did not enter the SBE Period) who were assigned to PF-06651600 in the Non-Responder Segment of the SBE Period
- Single Blind Extension-Active Non-responders on PF-06700841: Participants initially treated with PF-06700841 in the Initial 24-Week Treatment Period and not responsive at Week 24 (ie, not achieving SALT 30) who were continually assigned to PF-06700841 in the Non-Responder Segment of the SBE Period
- Single Blind Extension-Placebo Non-responders on PF-06700841: Participants initially treated with placebo in the Initial 24-Week Treatment Period who were assigned to PF-06700841 in the Non-Responder Segment of the SBE Period
- SBE-Non-Retreated PF-06651600 Responders in Withdrawal Segment: Participants initially treated with PF-06651600 in the Initial 24-Week Treatment Period and responsive at Week 24 (ie, achieving SALT 30) who were assigned to placebo (withdrawal) without entering the Retreatment Segment of the SBE Period
- SBE-Retreated PF-06651600 Responders in Withdrawal Segment: Participants initially treated with PF-06651600 in the Initial 24- Week Treatment Period and responsive at Week 24 (ie, achieving SALT 30) who were assigned to placebo (withdrawal), and then entered the Retreatment Segment of the SBE Period to receive PF-06651600.
  This arm described AEs for retreated responders within withdrawal Segment.
- SBE-Non-Retreated PF-06700841 Responders (Withdrawal Segment): Participants initially treated with PF-06700841 in the Initial 24-Week Treatment Period and responsive at Week 24 (ie, achieving SALT 30) who were assigned to placebo (withdrawal) without entering the Retreatment Segment of the SBE Period
- SBE-Retreated PF-06700841 Responders in the Withdrawal Segment: Participants initially treated with PF06700841 in the Initial 24- Week Treatment Period and responsive at Week 24 (ie, achieving SALT 30) who were assigned to placebo (withdrawal), and then entered the Retreatment Segment of the SBE Period to receive PF-06700841.This arm described AEs for retreated responders within Withdrawal Segment
- SBE-Retreated PF-06651600 Responders in Retreatment Segment: Participants initially treated with PF-06651600 in the Initial 24-Week Treatment Period and responsive at Week 24 (ie, achieving SALT 30) who were assigned to placebo (withdrawal), and then entered the Retreatment Segment of the SBE Period to receive PF-06651600
- SBE-Retreated Responders on PF-06700841 in Retreatment Segment: Participants initially treated with PF-06700841 in the Initial 24-Week Treatment Period and responsive at Week 24 (ie, achieving SALT 30) who were assigned to placebo (withdrawal), and then entered the Retreatment Segment of the SBE Period to receive PF-06700841
- Cross Over Extension-PF-06651600: Participants not responsive to placebo or PF-06700841 at Week 24 in the Initial 24-Week Treatment Period and not responsive to PF-06700841 at Week 52 (ie, not achieving SALT 30) in the SBE Period who were assigned to PF-06651600 in the COE Period
- Cross Over Extension-PF-06700841: Participants not responsive to placebo or PF-06651600 at Week 24 in the Initial 24-Week Treatment Period and not responsive to PF-06651600 at Week 52 (ie, not achieving SALT 30; except 1 PF-06651600 responder) in the SBE Period who were assigned to PF-06700841 in the COE Period
Arm/Group | Treatment Period-Placebo | Treatment Period-PF-06651600 | Treatment Period-PF-06700841 | Single Blind Extension-Active Non-responders on PF-06651600 | Single Blind Extension-Placebo Non-responders on PF-06651600 | Single Blind Extension-Active Non-responders on PF-06700841 | Single Blind Extension-Placebo Non-responders on PF-06700841 | SBE-Non-Retreated PF-06651600 Responders in Withdrawal Segment | SBE-Retreated PF-06651600 Responders in Withdrawal Segment | SBE-Non-Retreated PF-06700841 Responders (Withdrawal Segment) | SBE-Retreated PF-06700841 Responders in the Withdrawal Segment | SBE-Retreated PF-06651600 Responders in Retreatment Segment | SBE-Retreated Responders on PF-06700841 in Retreatment Segment | Cross Over Extension-PF-06651600 | Cross Over Extension-PF-06700841
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48 | 0/47 | 0/16 | 0/17 | 0/5 | 0/12 | 0/8 | 0/14 | 0/9 | 0/14 | 0/14 | 0/15 | 0/5 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48 | 2/47 | 0/16 | 0/17 | 0/5 | 0/12 | 0/8 | 0/14 | 0/9 | 0/14 | 0/14 | 1/15 | 0/5 | 1/18
Other Adverse Events (participants affected / at risk) | 26/47 | 23/48 | 28/47 | 8/16 | 12/17 | 4/5 | 10/12 | 4/8 | 3/14 | 6/9 | 9/14 | 11/14 | 8/15 | 4/5 | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period-Placebo (N=47) | Treatment Period-PF-06651600 (N=48) | Treatment Period-PF-06700841 (N=47) | Single Blind Extension-Active Non-responders on PF-06651600 (N=16) | Single Blind Extension-Placebo Non-responders on PF-06651600 (N=17) | Single Blind Extension-Active Non-responders on PF-06700841 (N=5) | Single Blind Extension-Placebo Non-responders on PF-06700841 (N=12) | SBE-Non-Retreated PF-06651600 Responders in Withdrawal Segment (N=8) | SBE-Retreated PF-06651600 Responders in Withdrawal Segment (N=14) | SBE-Non-Retreated PF-06700841 Responders (Withdrawal Segment) (N=9) | SBE-Retreated PF-06700841 Responders in the Withdrawal Segment (N=14) | SBE-Retreated PF-06651600 Responders in Retreatment Segment (N=14) | SBE-Retreated Responders on PF-06700841 in Retreatment Segment (N=15) | Cross Over Extension-PF-06651600 (N=5) | Cross Over Extension-PF-06700841 (N=18)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period-Placebo (N=47) | Treatment Period-PF-06651600 (N=48) | Treatment Period-PF-06700841 (N=47) | Single Blind Extension-Active Non-responders on PF-06651600 (N=16) | Single Blind Extension-Placebo Non-responders on PF-06651600 (N=17) | Single Blind Extension-Active Non-responders on PF-06700841 (N=5) | Single Blind Extension-Placebo Non-responders on PF-06700841 (N=12) | SBE-Non-Retreated PF-06651600 Responders in Withdrawal Segment (N=8) | SBE-Retreated PF-06651600 Responders in Withdrawal Segment (N=14) | SBE-Non-Retreated PF-06700841 Responders (Withdrawal Segment) (N=9) | SBE-Retreated PF-06700841 Responders in the Withdrawal Segment (N=14) | SBE-Retreated PF-06651600 Responders in Retreatment Segment (N=14) | SBE-Retreated Responders on PF-06700841 in Retreatment Segment (N=15) | Cross Over Extension-PF-06651600 (N=5) | Cross Over Extension-PF-06700841 (N=18)
Acne (Skin and subcutaneous tissue disorders) | 2 | 5 | 5 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Papulopustular rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
IgA nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 5 | 6 | 4 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 6 | 6 | 4 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 3 | 1 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 11 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lip oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelids pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bartholin's abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT02974868/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT02974868/SAP_001.pdf